CLINICAL TRIAL: NCT05753982
Title: Infuence of Kinesiotaping on Pulmonary Function Improvement in Multiple Rib Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Marko Zlicar, Principal Investigator, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Kinesiotape_RT
Record Dates: First submitted 2023-02-22; First posted 2023-03-03 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Chest Wall Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- kinesiotape (Experimental): Placement of kinesiotapes, using ligament techniques on the injured side of chest, focusing on the point of maximal pain.
  Interventions: Other: Kinesiotape placement
- control (Placebo Comparator): No kinesiotape, standard of care
  Interventions: Other: Kinesiotape placement

INTERVENTIONS:
Other: Kinesiotape placement — Placement of kinesiotapes, using ligament techniques on the injured side of chest, focusing on the point of maximal pain.

SUMMARY:
Elastic tapes, named "kinesiotapes" have a limited, but proven influence on pain reduction, improvement in muscular strength and joint function. It can be hypothetised that by using kinesiotape techniques on damaged chest wall (due to mostly rib fracture) we can improve not only analgesia, but also improve lung function tests and speed recovery.

DETAILED DESCRIPTION:
Chest wall injury changes the function of chest wall muscles and other structures, which in turn influences respiratory function and cause significant pain.

Elastic tapes, named "kinesiotapes" have a limited, but proven influence on pain reduction, improvement in muscular strength and joint function. It can be hypothetised that by using kinesiotape techniques on damaged chest wall (due to mostly rib fracture) we can improve not only analgesia, but also improve lung function tests and speed recovery.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral chest wall injury with multiple rib fracture (< 5 ribs)
* Signed informed consent

Exclusion Criteria:

* Minors
* Pregnant women
* Contraindications of using kinesiotapes
* Contraindications to perform spirometry (lung function tests)
* Inability to cooperate
* Chest drains
* Pneumothorax

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-08-27 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Improved spirometry tests | 2 days
  Improvement in lung function using spirometry

SECONDARY OUTCOMES:
Reduction in opioid consumption | 2 days
  Reduction in consumtion of opioid analgetic drugs

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No